CLINICAL TRIAL: NCT03218098
Title: Post-Operative Pain After Uniportal Vats Lobectomy: Does A Smaller Incision Result In Better Recovery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mohsen Ibrahim, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1037/2012
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Smaller Incision (Experimental): UVATS access for lobectomy with small skin access 4 cm
  Interventions: Procedure: Lobectomy via UVATS
- Traditional Incision (Active Comparator): UVATS access for lobectomy with longer skin access 8 cm
  Interventions: Procedure: Lobectomy via UVATS

INTERVENTIONS:
Procedure: Lobectomy via UVATS — lobectomy with small skin access 4 cm

SUMMARY:
Post-Operative Pain After Uniportal Vats Lobectomy: Does A Smaller Incision Result In Better Recovery?

Postoperative pain control remains one of the most common problems after major lung resection. Pain is considered a major independent factor responsible for increased perioperative morbidity and mortality: in particular, in patients with preoperative compromised clinical conditions. In fact, acute pain may compromise the patient's mobilization and the secretion's clearance with secondary possible bronchial obstruction and parenchymal lung infection.

Today, the treatment of postoperative pain after lung resection is based on association of the pharmacological therapy, including systemic use of opioids and non-steroid drugs, epidural analgesia, intercostal nerve block and cryoanalgesia with the minimally invasive surgery, like use of mini-thoracotomy, a thoracoscopic approach or intercostal nerve protection with the use of muscle sparing. In the literature, reduced tissue damage consequent to the use of limited surgical approaches is reported to be significantly effective in decreasing early postoperative pain. Thus, the use of a minimally invasive surgery for lung resections has proved to produce more tolerable pain and allow quicker functional recovery and lower postoperative complications. The aim of this prospective randomized study was to evaluate the equivalency of a smaller incision (4 cm) when compared to a longer length (8 cm) of incision performing uniportal VATS lobectomy in terms of postoperative pain results. Primarily, to evaluate the differences of operative time between the groups.

Secondly, to investigate the differences of pain scores between the two groups and the impact of pain reduction on functional results.

ELIGIBILITY:
Inclusion Criteria:

* be aged ≥ 18 years (of either gender)
* have provided written informed consent prior to participation in the study
* undergoing to major lung surgery with an Uniportal VideoThoracocopic Access (UVATS).

Exclusion Criteria:

* rethoracotomy
* presence of pleural adhesions
* Neuropathy
* be a participant in another interventional clinical trial or have received another investigational device or device within the last 30 days (donation of excised tissue [lung or parts of lymph nodes] for biological research may occur in the same patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Operative time reduction | up to 180 min
  Operative time reduction in minutes

SECONDARY OUTCOMES:
pain score | up to 48 hours
  VAS score